CLINICAL TRIAL: NCT07173868
Title: A Prospective Cohort Study Comparing Metabolic Response Evaluation by F-18 FDG PET-CT Versus Conventional Imaging for Outcome Stratification in Patients With Advanced Breast Cancer Receiving First-line Systemic Therapy
Brief Title: FDG PET-CT in Advanced Breast Cancer
Acronym: PET-000
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, Clinical Professor, Samsung Medical Center
Other Study IDs: 2025-06-039
Record Dates: First submitted 2025-08-20; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Histologically Confirmed Metastatic or Locally Advanced Breast Cancer With no Radical Topical Treatment Available; If There is Liver Metastasis, Which the Researcher Believes Will be Difficult to Evaluate the Response Accurately With Bone Metastasis or CT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- F-18 FDG PET-CT in advanced breast cancer: histologically confirmed metastatic or locally advanced breast cancer with no radical topical treatment available
  If there is liver metastasis, which the researcher believes will be difficult to evaluate the response accurately with bone metastasis or CT

SUMMARY:
This study is a prospective cohort study comparing metabolic response evaluation by F-18 FDG PET-CT versus conventional imaging for outcome stratification in patients with advanced breast cancer receiving first-line systemic therapy.

DETAILED DESCRIPTION:
PET-CT, CE-CT ± bone scan are performed before and during treatment (6, 12, 24, 48 weeks) of the first systemic treatment in a total of 100 patients with advanced breast cancer, and some patients analyze ctDNA-based MRD by collecting blood at the same time point. We analyze the relationship between patient-specific responses and PFS, and compare the predictive performance of imaging and molecular indicators.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years of age or older
2. histologically confirmed metastatic or locally advanced breast cancer with no radical topical treatment available
3. If there is liver metastasis, which the researcher believes will be difficult to evaluate the response accurately with bone metastasis or CT
4. May or may not have measurable lesions in accordance with RECIST 1.1 criteria
5. Patients who meet the criteria for coverage of F-18 FDG PET-CT tests conducted for the purpose of evaluating treatment response according to the Health Insurance Review and Assessment Service's announcement
6. Patients scheduled to start primary systemic therapy for advanced breast cancer (endocrine therapy, targeted therapy, chemotherapy, immunotherapy or their combination therapy)
7. Patients willing to undergo continuous response assessments using F-18 FDG PET-CT and CE-CT (± bone scan if clinically necessary) at the time point specified in the study plan (before treatment, 6, 12, 24, 48 weeks after treatment) and willing to pay for the examination accordingly
8. ECOG Performance Status 0-2

Exclusion Criteria:

1. a patient who has previously received systemic treatment for advanced breast cancer
2. Taboos for F-18 FDG PET-CT (e.g., uncontrolled diabetes) or intravenous contrast agents for CE-CT (e.g., severe allergies, severe renal dysfunction)
3. Pregnancy or lactation
4. At the same time, other primary malignancies (except when treatment has been completed for radical purposes) are known
5. Other medical conditions that, at the discretion of the researcher, may hinder participation in the study or affect the interpretation of the results
6. If you are unable to follow a research procedure or follow-up

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed metastatic or locally advanced breast cancer patients with no radical topical treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Follow up the response for 48 weeks after the start of the first systemic treatment | Within 4 weeks prior to the start of primary systemic treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical Center, Seoul, Gannam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No